CLINICAL TRIAL: NCT04961359
Title: A Randomized, Blinded, Placebo-controlled Phase Ⅰ Clinical Trial of Recombinant New Coronavirus Vaccine (CHO Cells) in the Safety and Tolerability of Healthy People Aged 3 to 17 Years of Age
Brief Title: Recombinant New Coronavirus Vaccine (CHO Cells) to Prevent SARS-CoV-2（COVID-19） Phase I Clinical Trial (3~17 Years Old)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Anhui Zhifei Longcom Biologic Pharmacy Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LKM-2021-NCV01
Record Dates: First submitted 2021-07-08; First posted 2021-07-14 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Coronavirus
Keywords: Recombinant Novel Coronavirus Vaccine
MeSH Terms: conditions — Coronavirus Infections | interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Population Ⅰ (Experimental): Population Ⅰ has 20 subjects aged 12 to 17 and is considered negative for SARS-COV-2 and fluorescent RT-PCR nucleic acids. PopulationⅠis intramuscular injection of deltoid muscle of upper arm with vaccine.
  Interventions: Biological: Recombinant new coronavirus vaccine (CHO cell) group
- Population Ⅱ (Placebo Comparator): Population Ⅱ has 5 subjects aged 12 to 17 and is considered negative for SARS-COV-2 and fluorescent RT-PCR nucleic acids. Population Ⅱ is a placebo intramuscular injection of deltoid muscle of the upper arm.
  Interventions: Biological: Recombinant new coronavirus vaccine (CHO cells) placebo group
- Population Ⅲ (Experimental): Population Ⅲ has 20 subjects aged 6 to 11 and is considered negative for SARS-COV-2 and fluorescent RT-PCR nucleic acids. Population Ⅲ is intramuscular injection of deltoid muscle of upper arm with vaccine.
  Interventions: Biological: Recombinant new coronavirus vaccine (CHO cell) group
- Population Ⅳ (Placebo Comparator): Population Ⅳ has 5 subjects aged 6 to 11 and is considered negative for SARS-COV-2 and fluorescent RT-PCR nucleic acids. Population Ⅳ is a placebo intramuscular injection of deltoid muscle of the upper arm.
  Interventions: Biological: Recombinant new coronavirus vaccine (CHO cells) placebo group
- Population Ⅴ (Experimental): Population Ⅴ has 20 subjects aged 3 to 5 and is considered negative for SARS-COV-2 and fluorescent RT-PCR nucleic acids. PopulationⅤ is intramuscular injection of deltoid muscle of upper arm with vaccine.
  Interventions: Biological: Recombinant new coronavirus vaccine (CHO cell) group
- Population Ⅵ (Placebo Comparator): Population Ⅵ has 5 subjects aged 3 to 5 and is considered negative for SARS-COV-2 and fluorescent RT-PCR nucleic acids. Population Ⅵ is a placebo intramuscular injection of deltoid muscle of the upper arm.
  Interventions: Biological: Recombinant new coronavirus vaccine (CHO cells) placebo group

INTERVENTIONS:
Biological: Recombinant new coronavirus vaccine (CHO cell) group — Intramuscular injection of deltoid muscle of upper armof 25μg/0.5ml/person doseRecombinant new coronavirus vaccine (CHO cells).
  Arms: Population Ⅰ; Population Ⅲ; Population Ⅴ
Biological: Recombinant new coronavirus vaccine (CHO cells) placebo group — Intramuscular injection of deltoid muscle of upper armof 0.5ml/person doseRecombinant new coronavirus vaccine (CHO cells) placebo.
  Arms: Population Ⅱ; Population Ⅳ; Population Ⅵ

SUMMARY:
Popular topic: Phase I clinical trial of recombinant new coronavirus vaccine (CHO cell) (3~17 years old) Research purpose:Main purpose:To evaluate the safety and tolerability of recombinant New Coronavirus vaccine (CHO cells) in healthy people aged 3 to 17. Secondary purpose: To explore the immunogenicity and persistence of recombinant New Coronavirus vaccine (CHO cells) in healthy people aged 3 to 17.

Overall design:A single center, randomized, blind, placebo-controlled trial design was adopted.

Study population: 75 healthy people aged 3 to 17 years old, both male and female.

Test groups: 3 to 5 years old: 20 cases in experimental group and 5 cases in placebo group; 6 to 11 years old: 20 patients in the experimental group and 5 patients in the placebo group; 12 to 17 years old: 20 patients in experimental group and 5 patients in placebo group.

DETAILED DESCRIPTION:
Popular topic: Phase I clinical trial of recombinant new coronavirus vaccine (CHO cell) (3~17 years old) .

Product name: Recombinant new coronavirus vaccine (CHO cell),Each dose contains 25μgNCP-RBD protein/0.5mL/bottle.

Indications: Prevention of respiratory diseases caused by new coronavirus infection .

Research population: healthy people aged 3 to 17 . Research Unit: Hunan Provincial Center for Disease Control and Prevention. Research purpose:Main purpose:To evaluate the safety and tolerability of recombinant New Coronavirus vaccine (CHO cells) in healthy people aged 3 to 17. Secondary purpose: To explore the immunogenicity and persistence of recombinant New Coronavirus vaccine (CHO cells) in healthy people aged 3 to 17.

Overall design:A single center, randomized, blind, placebo-controlled trial design was adopted.

Immunization program: 0, 1, and 2 months. Dose:25μg/0.5mL/bottle. Study population: 75 healthy people aged 3 to 17 years old, both male and female.

Test groups: 3 to 5 years old: 20 cases in experimental group and 5 cases in placebo group; 6 to 11 years old: 20 patients in the experimental group and 5 patients in the placebo group; 12 to 17 years old: 20 patients in experimental group and 5 patients in placebo group.

Research plan and implementation:According to the age from big to small, it was divided into three stages: 12 to 17 years old, 6 to 11 years old, 3 to 5 years old. The subjects of each age group were randomly divided into the experimental vaccine group and the placebo control group, 20 in the experimental vaccine group and 5 in the placebo group.

In the first stage, the subjects aged 12 to 17 years old were randomly divided into the experimental vaccine group (20 cases) and the placebo group (5 cases); The safety data of 0-7 days after the first dose were evaluated by the researchers. If the suspension / termination criteria were not met, the second phase of the study was carried out, and the subjects aged 6-11 years old in the trial vaccine group (20 cases) and placebo group (5 cases) were randomly enrolled; The safety data of subjects aged 6 to 17 years old from 0 to 7 days after the second dose of vaccine were evaluated by the researchers. If the suspension / termination criteria were not met, the third phase study was carried out, and the subjects aged 3 to 5 years old in the trial vaccine group (20 cases) and placebo group (5 cases) were randomly enrolled.

The subjects were followed up for 30 days after each dose. If the suspension / termination criteria were met, DSMB would decide whether to vaccinate the next dose; In other cases, it was up to the researchers to decide whether or not to receive the follow-up dose.

Safety endpoint:

1. The incidence of all AEs within 1 month after the first dose to the full course of vaccination:

1. Total AE incidence;
2. The incidence of AEs related to research vaccines;
3. The incidence of grade 3 and above AE;
4. The incidence of grade 3 and above AEs related to research vaccines;
5. The incidence of AEs leading to withdrawal;
6. The incidence of AEs related to research vaccines leading to withdrawal; 2. The incidence of all serious adverse events (SAE) and the incidence of SAE related to the vaccine within 12 months after the first dose to the full course of vaccination; 3. Changes in the clinical significance of the laboratory test indicators after first and second dose of inoculation compared to before the first dose.

Immunogenicity endpoint:

Humoral immunity: before the first dose of vaccination, 1 month,3 month and 6 months after the full vaccination, neutralizing antibodies of novel coronavirus (SARS-CoV-2), S protein binding antibody (IgG), RBD protein binding antibody (IgG) ) Positive rate; The levels of neutralizing antibodies against SARS-CoV-2, S protein binding antibody (IgG) and RBD protein binding antibody (IgG) and their relative immunity 1 month , 3 month and 6 months after the full vaccination of all subjects increase the multiple before.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 3-17 years old (all inclusive);
2. The subject voluntarily agrees to participate in the study (or the legal guardian of the subject voluntarily agrees the child to participate in the study), and the guardian and the subject (8-17 years old) sign the informed consent form, and can provide valid identification; Understand and comply with test protocol requirements;
3. The subject and / or the legal guardian of the subject have the ability to understand the (non illiterate) study procedure and participate in the planned follow-up;
4. Axillary temperature < 37.3 ℃ (> 14 years old), axillary temperature < 37.5 ℃(≤14 years old);
5. Female and male subjects of childbearing age agreed to take effective contraceptive measures during the study.

Exclusion Criteria:

1. The results of physical examination and laboratory examination before screening were abnormal and clinically significant;
2. Any component of the test vaccine, including aluminum preparation, has a history of severe allergy, such as anaphylactic shock, allergic laryngeal edema, allergic purpura, thrombocytopenic purpura, local allergic necrosis reaction (Arthus reaction), dyspnea, angioneurotic edema, etc; Or the above-mentioned serious adverse reactions occurred after the use of any vaccine or drug in the past;
3. Patients with history of SARS and SARS-CoV-2 (meet any of the following items):

   ① History of infection or history of SARS and SARS-CoV-2;

   ② During the epidemic of sras-cov-2, there was a history of contact with patients diagnosed / suspected with new crown;

   ③ The detection of SARS-CoV-2 IgM and / or IgG antibody was positive;

   ④ RT-PCR was positive.
4. They had taken antipyretics or analgesics within 24 hours before the first dose of vaccine;
5. those who have been vaccinated with New Coronavirus or inoculated with live attenuated vaccine within 30 days within 14 days before the first dose of the vaccine are inoculated with the subunit vaccine and / or inactivated vaccine;
6. Patients with the following diseases:

   ① Patients with acute (within 72 hours) febrile diseases (> 14 years old, axillary temperature ≥ 37.3 ℃; ≤4 years old,axillary temperature ≥37.5 ℃);

   ② Digestive system diseases (such as diarrhea, abdominal pain, vomiting, etc.) in the past 7 days;

   ③ Suffering from congenital malformations or developmental disorders, genetic defects, severe malnutrition, etc;

   ④ A history of congenital or acquired immunodeficiency or autoimmune disease or immunomodulatory therapy within 6 months, such as immunosuppressive dose of glucocorticoid (dose reference: equivalent to prednisone 20mg / day, more than one week); or monoclonal antibody; or thymosin; or interferon, etc; however, local medication (such as ointment, eye drops, inhaler or nasal spray) is allowed;

   ⑤ Known to be diagnosed with infectious diseases, such as active tuberculosis, viral hepatitis, present or / or human immunodeficiency virus HIV antibody positive or syphilis specific antibody positive, or parents who are HIV infected;

   ⑥ Neurological diseases or neurodevelopmental disorders (e.g., migraine, epilepsy, stroke, seizures in the last three years, encephalopathy, focal neurological deficit, Guillain Barre syndrome, encephalomyelitis or transverse myelitis); History of mental illness or family history;

   ⑦ Functional asplenia and splenectomy for any reason;

   ⑧ There are serious chronic diseases or disease in progress can not be controlled smoothly, such as diabetes, thyroid disease;

   ⑨ Severe liver and kidney diseases; Current respiratory diseases requiring daily medication (e.g., chronic obstructive pulmonary disease [COPD], asthma) or any treatment for exacerbation of respiratory diseases (e.g., asthma exacerbation) in the last five years; A history of severe cardiovascular disease (such as congestive heart failure, cardiomyopathy, ischemic heart disease, arrhythmia, conduction block,myocardial infarction, pulmonary heart disease), or myocarditis or pericarditis;

   ⑩ Thrombocytopenia, any coagulation dysfunction or anticoagulant therapy, etc;

   ⑪ Cancer patients.
7. Received blood or blood related products, including immunoglobulin, within 3 months; or planned use during the study period;
8. Have been pregnant (including positive urine pregnancy test), or in lactation;
9. Use any research or unregistered product (drug, vaccine, biological product or device) other than the research product within 3 months, or plan to use it during the research period;
10. Researchers believe that any disease or condition of the subject may put the subject at an unacceptable risk; The subjects could not meet the requirements of the protocol; Interference with the assessment of vaccine response.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2021-07-03 (Actual); Primary Completion 2021-12-12 (Actual); Study Completion 2023-04-06 (Actual)

PRIMARY OUTCOMES:
The number of adverse events after intramuscular injection | 12 months after full vaccination
  The main observation methods of adverse reactions mainly include laboratory examination, local reactions and systemic reactions at the administration site.
Immunogenic end point | Within 6 months after the last dose of vaccination
  The positive rate of neutralizing antibody, S protein binding antibody (IgG), RBD protein binding antibody (IgG) of all subjects before the first dose, 1 month，3 months and 6 months after the full vaccination. And titer levels and their fold increase before immunity.

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Provincial Center for Disease Control and Prevention, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gao L, Li Y, He P, Chen Z, Yang H, Li F, Zhang S, Wang D, Wang G, Yang S, Gong L, Ding F, Ling M, Wang X, Ci L, Dai L, Gao GF, Huang T, Hu Z, Ying Z, Sun J, Zuo X. Safety and immunogenicity of a protein subunit COVID-19 vaccine (ZF2001) in healthy children and adolescents aged 3-17 years in China: a randomised, double-blind, placebo-controlled, phase 1 trial and an open-label, non-randomised, non-inferiority, phase 2 trial. Lancet Child Adolesc Health. 2023 Apr;7(4):269-279. doi: 10.1016/S2352-4642(22)00376-5. Epub 2023 Feb 17. PMID 36803632